CLINICAL TRIAL: NCT00254267
Title: An Open-label Phase 2 Study of AMG 706 in Japanese Subjects With Advanced Gastrointestinal Stromal Tumors (GISTs) Who Developed Progressive Disease or Relapsed While on Imatinib Mesylate
Brief Title: Evaluate the Efficacy of AMG 706 to Treat Advanced Gastrointestinal Stromal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050129
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Advanced Gastrointestinal Stromal Tumor
Keywords: Gastrointestinal Stromal Tumor, Imatinib Mesylate Resistance, Phase2 study, AMG 706
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — motesanib diphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm One (Experimental): AMG 706 125mg, oral, once a day
  Interventions: Drug: AMG 706

INTERVENTIONS:
Drug: AMG 706 — AMG 706 125mg, oral, once a day

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of AMG 706 in patients with gastrointestinal stromal tumor that have not been controlled while taking imatinib mesylate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histological confirmed GIST
* Had prior imatinib mesylate therapy
* Has at least 1 measurable leasion by modified RECIST

Exclusion Criteria:

* Central nervous system tumor involvement requiring treatment
* History of myocardial infraction
* Uncontrolled hypertension

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-11; Primary Completion 2007-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The objective response rate as assessed by modified RECIST | Every 8 weeks

SECONDARY OUTCOMES:
Duration of response, progression-free survival, time to response, overall survival, PK and safety profile | imaging, every 8 weeks; survival, every 6 months; PK, Days 1,15, 29, 43, 57, every 2 weeks in week 9 to 16, and every 4 weeks thereafter;

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Benjamin RS, Schoffski P, Hartmann JT, Van Oosterom A, Bui BN, Duyster J, Schuetze S, Blay JY, Reichardt P, Rosen LS, Skubitz K, McCoy S, Sun YN, Stepan DE, Baker L. Efficacy and safety of motesanib, an oral inhibitor of VEGF, PDGF, and Kit receptors, in patients with imatinib-resistant gastrointestinal stromal tumors. Cancer Chemother Pharmacol. 2011 Jul;68(1):69-77. doi: 10.1007/s00280-010-1431-9. Epub 2010 Sep 14. PMID 20838998
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com